CLINICAL TRIAL: NCT05567926
Title: Acute Effects of Beetroot Juice Ingestion on Isometric Knee Extension Strength, Explosive Strength and Local Muscular Endurance
Brief Title: Acute Effects of Beetroot Juice on Isometric Knee Extension Strength, Explosive Strength and Local Muscular Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate Professor, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BEETROOT
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Healthy Adults
Keywords: isometric strength; beetroot; nitrates; local muscle endurance; supplementation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition, receiving beetroot juice supplement (Experimental): Participants will receive beetroot juice intervention in the experimental condition.
  Interventions: Dietary Supplement: Beetroot juice concentrate (140 ml)
- Placebo condition (Placebo Comparator): Participants will receive placebo (blackcurrant juice) in the placebo condition
  Interventions: Dietary Supplement: Blackcurrant juice (placebo)

INTERVENTIONS:
Dietary Supplement: Beetroot juice concentrate (140 ml) — A beetroot juice concentrate (140 ml) will be administered to participants in experimental conditions.
  Arms: Experimental condition, receiving beetroot juice supplement
Dietary Supplement: Blackcurrant juice (placebo) — 140 ml of blackcurrant juice with added appropriate amount of sugar to equalize the carbohydrate value and lemon juice fort the taste.
  Arms: Placebo condition

SUMMARY:
This is a double-blind placebo-controlled cross-over trial that aims to determine the acute effect of beetroot juice ingestion on isometric knee extension strength, explosive strength and local muscular endurance.

DETAILED DESCRIPTION:
The study aims to determine whether concentrated beetroot juice has an acute effect on isometric strength of the knee muscles and the rate of force development in knee extension, as well as endurance of the same muscle. This will be a cross-over study. 20 subjects will be randomly selected to the experimental group or control group; after 1 week, participants will repeat the measurements in the other condition. Subjects will consume 140 ml of beetroot juice extract 2.5 hours before the measurement or placebo (140 ml of blackcurrant juice with added appropriate amount of sugar to equalize the carbohydrate value and lemon juice fort the taste). An isometric dynamometer will be used to measure the isometric strength of the knee extensors. Investigators will quantify peak force, rate of force development, endurance of knee extensors at 50 % of the maximal force, and the force recovery after a fatiguing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* Physically active and healthy athletes (recreational or professional)

Exclusion Criteria:

* Cardiovascular, pulmonary, metabolic, neurological diseases and musculoskeletal injuries
* Smokers
* Consumption of drugs such as antacids and proton pump inhibitors in the previous 3 months
* Pregnant or breastfeeding women
* Beetroot allergic participants

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Knee extension strength | 2 hours after the ingestion of beetroot juice or placebo
  The peak force during maximal voluntary contraction of knee extensors

SECONDARY OUTCOMES:
Knee extension explosive strength | 2 hours after the ingestion of beetroot juice or placebo
  The rate of force development during maximal voluntary contraction of knee extensors
Knee extension local muscle endurance | 2 hours after the ingestion of beetroot juice or placebo
  Time to failure of knee muscles at 50 % of maximal force

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided